CLINICAL TRIAL: NCT02631473
Title: Pharmacokinetics of Efavirenz and Lopinavir Nano-formulations in HIV Negative Healthy Volunteers: an Adaptive Design Study
Brief Title: PK of Efavirenz & Lopinavir Nano-formulations in Healthy Volunteers
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Study is on hold whilst a grant application for further funding is put together
Sponsor: St Stephens Aids Trust (Other)
Collaborators: University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSAT 055
Record Dates: First submitted 2015-01-06; First posted 2015-12-16 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: HIV
MeSH Terms: interventions — efavirenz; Ritonavir; lopinavir-ritonavir drug combination; Lopinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1st Stage-Group A (Active Comparator): 1. Day 1: 50 mg NANO-efavirenz single dose
  2. Days 4-21: 50 mg NANO-efavirenz OD (once daily)
  Interventions: Drug: 50mg NANO-efavirenz
- 1st Stage-Group B (Active Comparator): 1. Days 1-7: 400mg NANO-lopinavir BID (twice daily)
  2. Days 8-21: Wash-out period
  3. Days: 22-28: 200mg NANO-lopinavir BID plus 100mg Ritonavir (Norvir) BID
  Interventions: Drug: 400mg NANO-Lopinavir; Drug: 200mg NANO-Lopinavir; Drug: 100mg Ritonavir
- 2nd Stage-Group A-Group 1-Dose level 1 (Active Comparator): 1. 21 Days: 300mg NANO-efavirenz OD
  2. 4 weeks: Wash-out period
  3. 21 days: 600mg Sustiva OD
  Interventions: Drug: 300mg NANO-Efavirenz; Drug: 600mg Sustiva
- 2nd Stage-Group A-Group 2-Dose level 2 (Active Comparator): 1. 21 Days: 200mg NANO-efavirenz OD
  2. 4 weeks: Wash-out period
  3. 21 days: 400mg Sustiva OD
  Interventions: Drug: 200mg NANO-Efavirenz; Drug: 400mg Sustiva
- 2nd Stage-Group B-Arm 1 (Active Comparator): 1. 7 days: Kaletra® (lopinavir400mg/ritonavir100mg) BD
  2. 2 weeks: Wash-out period
  3. 7 days: NANO-lopinavir (200mg +/- ritonavir®)
  Interventions: Drug: Kaletra® (lopinavir 400mg/ritonavir 100mg); Drug: +/- 200mg NANO-Lopinavir; Drug: +/- 200mg ritonavir NORVIR
- 2nd Stage-Group B-Arm 2 (Active Comparator): 1. 7 days: NANO-lopinavir (200mg +/- ritonavir Norvir)
  2. 2 weeks: Wash-out period
  3. 7 days: Kaletra® (lopinavir400mg/ritonavir100mg) BD
  Interventions: Drug: Kaletra® (lopinavir 400mg/ritonavir 100mg); Drug: +/- 200mg NANO-Lopinavir; Drug: +/- 200mg ritonavir NORVIR

INTERVENTIONS:
Drug: 50mg NANO-efavirenz — OD
  Arms: 1st Stage-Group A
Drug: 400mg NANO-Lopinavir — BID
  Arms: 1st Stage-Group B
Drug: 200mg NANO-Lopinavir — BID
  Other Names: Efavirenz
  Arms: 1st Stage-Group B
Drug: 100mg Ritonavir — BID
  Other Names: Norvir
  Arms: 1st Stage-Group B
Drug: 300mg NANO-Efavirenz — OD
  Arms: 2nd Stage-Group A-Group 1-Dose level 1
Drug: 600mg Sustiva — OD
  Other Names: Efavirenz
  Arms: 2nd Stage-Group A-Group 1-Dose level 1
Drug: 200mg NANO-Efavirenz — OD
  Arms: 2nd Stage-Group A-Group 2-Dose level 2
Drug: Kaletra® (lopinavir 400mg/ritonavir 100mg) — BID
  Other Names: Lopinavir/Ritonavir
  Arms: 2nd Stage-Group B-Arm 1; 2nd Stage-Group B-Arm 2
Drug: +/- 200mg NANO-Lopinavir — BID
  Arms: 2nd Stage-Group B-Arm 1; 2nd Stage-Group B-Arm 2
Drug: +/- 200mg ritonavir NORVIR — BID
  Other Names: Ritonavir
  Arms: 2nd Stage-Group B-Arm 1; 2nd Stage-Group B-Arm 2
Drug: 400mg Sustiva
  Other Names: Efavirenz
  Arms: 2nd Stage-Group A-Group 2-Dose level 2

SUMMARY:
This study is an open-label, prospective pharmacokinetic study investigating two antiretroviral agents in parallel and employing an adaptive design with two stages, whereby the results obtained in the primary stage inform the doses selected for investigation in the secondary stage

DETAILED DESCRIPTION:
The objectives of this study are:

Primary

* To investigate the pharmacokinetics of a new pharmaceutical formulation of efavirenz (NANO-efavirenz) in HIV negative healthy volunteers after single dose and a steady-state.
* To investigate the pharmacokinetics of a new pharmaceutical formulation of lopinavir (NANO-lopinavir) in HIV negative healthy volunteers

Secondary

* To investigate the safety and tolerability of NANO-efavirenz and NANO-lopinavir in HIV negative healthy volunteers
* To assess the bioequivalence of a selected single-dose of NANO-efavirenz to a single dose 600mg of efavirenz as Sustiva®
* To investigate the association between genetic polymorphisms in drug disposition genes and drug exposure

ELIGIBILITY:
Inclusion Criteria:

Volunteers must meet all of the following inclusion criteria within 28 days prior to the baseline visit:

1. The ability to understand and sign a written informed consent form, prior to participation in any screening procedures and must be willing to comply with all study requirements
2. Male or non-pregnant, non-lactating females
3. Between 18 to 65 years, inclusive
4. Body Mass Index (BMI) of 18 to 30 kg/m2, inclusive
5. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for a period of at least 12 weeks after the study

   A female may be eligible to enter and participate in the study if she:
   1. is of non-child-bearing potential defined as either post-menopausal (12 months of spontaneous amenorrhea and ≥ 45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy or,
   2. is of child-bearing potential with a negative pregnancy test at both Screening and Day 1 and agrees to use one of the following methods of contraception to avoid pregnancy:

      * Complete abstinence from penile-vaginal intercourse from 2 weeks prior to administration of IP, throughout the study, and for at least 2 weeks after discontinuation of all study medications;
      * Double barrier method (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide);
      * Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year (not all IUDs meet this criterion, see protocol appendix 7 for an example listing of approved IUDs);
      * Condom and depot medroxyprogesterone acetate ( DMPA) injections
      * Male partner sterilization confirmed prior to the female subject's entry into the study, and this male is the sole partner for that subject;
      * Any other method with published data showing that the expected failure rate is <1% per year.
      * Any contraception method must be used consistently, in accordance with the approved product label and for at least 2 weeks after discontinuation of IP.
6. Willing to consent to their personal details being entered onto the TOPS database
7. Willing to provide proof of identity by photographic ID at screen and any subsequent visit
8. Registered with a GP in the UK

Exclusion Criteria:

Volunteers who meet any of the following exclusion criteria are not to be enrolled in this study.

1. Any significant acute or chronic medical illness including hypertension (BP persistently >140/90 mmHg) or hypotension (BP persistently <90/60 mmHg)
2. Prolongation of ECG intervals: PR > 200 msec or QTcF > 450 msec.
3. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations.
4. Liver transaminase (ALT or AST > 1.25 x the upper limit of the normal range)
5. Significant psychiatric history (including severe depression) or history of seizures.
6. Positive blood screen for either hepatitis B surface antigen or hepatitis C antibody
7. Positive blood screen for HIV-1 and/or 2 antibodies
8. Current or recent (within 3 months) gastrointestinal disease
9. Clinically relevant alcohol or drug use (positive urine drug screen) or history of alcohol or drug use considered by the Investigator to be sufficient to hinder adherence to treatment, follow-up procedures or evaluation of adverse events. Smoking is permitted, but tobacco intake should remain consistent throughout the study
10. Known cardiac disease history of any family history of sudden cardiac death.
11. Exposure to any investigational drug or placebo within 3 months of first dose of study drug
12. Use of any other drugs (unless approved by the Investigator), including over-the-counter medications and herbal preparations, within two weeks prior to first dose of study drug, unless approved/prescribed by the Principal Investigator as known not to interact with study drugs.
13. Females of childbearing potential without the use of effective non-hormonal birth control methods, or not willing to continue practising these birth control methods for at least 12 weeks after the end of the treatment period
14. Previous allergy to any of the constituents of the pharmaceuticals administered in this trial
15. Rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucosegalactose malabsorption

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
The pharmacokinetics of a new pharmaceutical formulation of efavirenz (NANOefavirenz) and lopinavir (NANOlopinavir) in HIV negative healthy volunteers, as measured by Ctrough | Assessed from baseline visit (day 1) to : 1) Day 31 (Primary Stage Group A); 2) Day 30 (Primary Stage Group B); 3) Day 80 (Secondary Stage Group A); 4) Day 30 (Secondary Stage Group B)
  Trough concentration (Ctrough) is defined as the concentration at 24 hours after the observed drug dose.
The pharmacokinetics of a new pharmaceutical formulation of efavirenz (NANOefavirenz) and lopinavir (NANOlopinavir) in HIV negative healthy volunteers, as measured by Cmax | Assessed from baseline visit (day 1) to : 1) Day 31 (Primary Stage Group A); 2) Day 30 (Primary Stage Group B); 3) Day 80 (Secondary Stage Group A); 4) Day 30 (Secondary Stage Group B)
  Cmax is defined as the maximum observed plasma concentration
The pharmacokinetics of a new pharmaceutical formulation of efavirenz (NANOefavirenz) and lopinavir (NANOlopinavir) in HIV negative healthy volunteers, as measured by t1/2 | Assessed from baseline visit (day 1) to : 1) Day 31 (Primary Stage Group A); 2) Day 30 (Primary Stage Group B); 3) Day 80 (Secondary Stage Group A); 4) Day 30 (Secondary Stage Group B)
  t1/2 is defined as the elimination half-life
The pharmacokinetics of a new pharmaceutical formulation of efavirenz (NANOefavirenz) and lopinavir (NANOlopinavir) in HIV negative healthy volunteers, as measured by Tmax | Assessed from baseline visit (day 1) to : 1) Day 31 (Primary Stage Group A); 2) Day 30 (Primary Stage Group B); 3) Day 80 (Secondary Stage Group A); 4) Day 30 (Secondary Stage Group B)
  Tmax is defined as the time point at Cmax (Tmax)
The pharmacokinetics of a new pharmaceutical formulation of efavirenz (NANOefavirenz) and lopinavir (NANOlopinavir) in HIV negative healthy volunteers, as measured by total drug exposure | Assessed from baseline visit (day 1) to : 1) Day 31 (Primary Stage Group A); 2) Day 30 (Primary Stage Group B); 3) Day 80 (Secondary Stage Group A); 4) Day 30 (Secondary Stage Group B)
  Total drug exposure will be expressed as the area under the plasma concentration-time curve (AUC): from 0-12 (AUC0-12h) and 0-56 hours (AUC0-56h) for lopinavir; or 0-24 (AUC0-24h) and 0-228 hours (AUC0-24h) for efavirenz.

SECONDARY OUTCOMES:
Safety and tolerability of NANOefavirenz and NANOlopinavir in HIV negative healthy volunteers, as measured by concomitant medication check | 1) From screening visit to day 45 (Primary Stage Group A); 2) From screening visit to day 44 (Primary Stage Group B); 3) From screening visit to day 94 (Secondary Stage Group A); 4) From screening visit to day 44 (Secondary Stage Group B)
Safety and tolerability of NANOefavirenz and NANOlopinavir in HIV negative healthy volunteers, as measured by Adverse Events | 1) From screening visit to day 45 (Primary Stage Group A); 2) From screening visit to day 44 (Primary Stage Group B); 3) From screening visit to day 94 (Secondary Stage Group A); 4) From screening visit to day 44 (Secondary Stage Group B)
Safety and tolerability of NANOefavirenz and NANOlopinavir in HIV negative healthy volunteers, as measured by symptom directed physical exam | 1) From screening visit to day 45 (Primary Stage Group A); 2) From screening visit to day 44 (Primary Stage Group B); 3) From screening visit to day 94 (Secondary Stage Group A); 4) From screening visit to day 44 (Secondary Stage Group B)
Safety and tolerability of NANOefavirenz and NANOlopinavir in HIV negative healthy volunteers, as measured by vital signs | 1) From screening visit to day 45 (Primary Stage Group A); 2) From screening visit to day 44 (Primary Stage Group B); 3) From screening visit to day 94 (Secondary Stage Group A); 4) From screening visit to day 44 (Secondary Stage Group B)
  Temperature, blood pressure, heart rate, and respiratory rate
Safety and tolerability of NANOefavirenz and NANOlopinavir in HIV negative healthy volunteers, as measured by ECG | 1) From screening visit to day 21 (Primary Stage Group A); 2) From screening visit to day 28 (Primary Stage Group B); 3) From screening visit to day 70 (Secondary Stage Group A); 4) From screening visit to day 28 (Secondary Stage Group B)
  12 lead ECG with calculation of corrected QT interval (Fredericia)
Safety and tolerability of NANOefavirenz and NANOlopinavir in HIV negative healthy volunteers, as measured by Urinalysis | ) From screening visit to day 21 (Primary Stage Group A); 2) From screening visit to day 28 (Primary Stage Group B); 3) From screening visit to day 70 (Secondary Stage Group A); 4) From screening visit to day 28 (Secondary Stage Group B)
  Glucose, ketones, blood, pH, proteins, nitrites and leucocytes Pregnancy test for females of childbearing potential (urine) Drug screen
Safety and tolerability of NANOefavirenz and NANOlopinavir in HIV negative healthy volunteers, as measured haematology | 1) From screening visit to day 45 (Primary Stage Group A); 2) From screening visit to day 44 (Primary Stage Group B); 3) From screening visit to day 94 (Secondary Stage Group A); 4) From screening visit to day 44 (Secondary Stage Group B)
  1. Coulter count with differential
  2. Clotting screen; PT, APTT, Fibrinogen
Safety and tolerability of NANOefavirenz and NANOlopinavir in HIV negative healthy volunteers, as measured by clinical chemistry | 1) From screening visit to day 45 (Primary Stage Group A); 2) From screening visit to day 44 (Primary Stage Group B); 3) From screening visit to day 94 (Secondary Stage Group A); 4) From screening visit to day 44 (Secondary Stage Group B)
  Serum Biochemistry - Including sodium, potassium, urea, creatinine, total cholesterol and triglycerides, calcium, phosphate, liver enzymes (ALT, AST, GGT), albumin, glucose.
Safety and tolerability of NANOefavirenz and NANOlopinavir in HIV negative healthy volunteers, as measured by Adherence questioning/ pill count | 1) Days 14 and 21 (Primary Stage Group A); 2) Days 7 and 28 (Primary Stage Group B); 3) Days 14, 21, 63, and 70 (Secondary Stage Group A); 4) Days 7 and 28 (Secondary Stage Group B)
Safety and tolerability of NANOefavirenz in HIV negative healthy volunteers, as measured by CNS symptoms questionnaire | 1) Days 2 and 21 (Primary Stage Group A); 2) Days 2, 21, 51, and 70 (Secondary Stage Group A)
Relationship between genetic polymorphisms and exposure to the studied drugs. | Sample taken at baseline (if consented)
  Preliminary comparison between genotype and phenotype

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, Principal Investigator — Chelsea & Westminster Hospital; Steve Rannard, Study Director — University of Liverpool
Locations (1):
- St Stephen's Centre, London, London, United Kingdom